CLINICAL TRIAL: NCT07143045
Title: A Prospective Cohort Study of Zorifertinib as a First-line Treatment in Patients With Epidermal Growth Factor Receptor-mutant Advanced Non-small Cell Lung Cancer With Central Nervous System (CNS) Metastases
Status: Recruiting | Type: Observational
Sponsor: Alpha Biopharma (Jiangsu) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: AZD3759-CIT-401
Record Dates: First submitted 2025-08-06; First posted 2025-08-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: EGFR Mutant Advanced Non-small Cell Lung Cancer; Central Nervous System (CNS) Metastases
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: Patients who receive first-line zorifertinib and meet the inclusion/exclusion criteria of the EVEREST study (the EVEREST study is a randomized, open-label, multi-center, Phase II/III study to compare the efficacy and safety of first-line zorifertinib versus gefitinib/erlotinib in EGFR-mutant advanced NSCLC patients with CNS metastases)
  Interventions: Drug: zorifertinib
- Cohort B: Patients who receive first-line zorifertinib but do not meet the inclusion/exclusion criteria of the EVEREST study (the EVEREST study is a randomized, open-label, multi-center, Phase II/III study to compare the efficacy and safety of first-line zorifertinib versus gefitinib/erlotinib in EGFR-mutant advanced NSCLC patients with CNS metastases)
  Interventions: Drug: zorifertinib
- Cohort C: Patients who receive various other anti-tumor drugs selected by the clinician, excluding zorifertinib, as first-line treatment.

INTERVENTIONS:
Drug: zorifertinib — Cohort A and B will receive zorifertinib as first line treatment
  Groups: Cohort A; Cohort B

SUMMARY:
This study is a patient-centered, two-group, three-cohort, multi-center, prospective study to further evaluate the survival benefits and safety of zorifertinib as a first-line treatment in EGFRm+ advanced NSCLC patients with CNS metastases, and to compare the clinical value of zorifertinib with other epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs).

ELIGIBILITY:
Inclusion criteria:

1. Male or female, aged ≥18 years.
2. Histologically or cytologically confirmed NSCLC with EGFR sensitizing mutations (including L858R or Exon 19Del), ineligible for curative surgery or radiotherapy.
3. CNS metastases diagnosed as brain metastases (BM) and/or leptomeningeal metastases (LM) by imaging and/or cerebrospinal fluid pathological examination.
4. Planning to receive zorifertinib (zorifertinib group) or other anti-tumor treatments (other treatment group) as first-line treatment.
5. Voluntarily agreeing to participate in this study and signing the informed consent form.

Exclusion criteria:

1. Currently participating or planning to participate in any interventional clinical study for first-line treatment (patients who have participated in non-interventional, real-world studies may still be included).
2. Other reasons that, in the Investigator's opinion, make the patient unsuitable for this study.

For patients in Cohort A of the zorifertinib group, the following inclusion/exclusion criteria of the EVEREST study must also be met:

Inclusion Criteria A:

1. . No prior treatment with chemotherapy, EGFR-TKIs, biological therapy, immunotherapy, or any investigational drug that is considered first line treatment for advanced NSCLC.
2. . Eligible patients are not candidates for definitive surgical resection or radiation of all lesions in the opinion of the treating physician.
3. . All patients must be stable without any systemic (oral or parenteral) corticosteroid or anticonvulsant therapy for at least 2 weeks prior to study treatment. Inhaled non-absorbable and topical corticosteroid use are permitted as indicated.
4. . Patients may have prior placement of a properly functioning CNS shunt or Ommaya reservoir.
5. . ECOG performance status 0 or 1, with no deterioration over the past 2 weeks, and expected survival time ≥ 3 months.
6. . Women of child-bearing potential (WOCBP) and male patients should agree to take medically acceptable contraception measures while on study treatment and for 3 months following completion of study treatment. All WOCBP must have a negative pregnancy test at screening.
7. . Patients with measurable CNS lesions must have at least one site of CNS lesion, which has not been previously irradiated, can be accurately measured at baseline as ≥ 10 mm in the longest diameter by MRI, and is suitable for accurate repeated measurements. Measurable extracranial lesions are not required. Patients with non-measurable CNS lesions must have at least one extracranial lesion, which has not been previously irradiated, can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except for lymph nodes which must have a short diameter ≥ 15 mm) by CT/MRI, and is suitable for accurate repeated measurements.

Exclusion Criteria A:

1. . Prior treatment with EGFR-TKIs (if EGFR-TKIs were used as adjuvant therapy, patients may be enrolled if the time from discontinuation to relapse meets the following requirements: >6 months for Cohort A, and >3 months for Cohorts B and C).
2. . Positive for T790M mutation documented by central or local laboratory using an approved or validated test method, or documented positive KRAS or cMET.
3. . Patients who have received any investigational drug, biological therapy, or immunotherapy for their malignant tumors within the past 21 days.
4. . Patients who have had a major surgical procedure (excluding the need for placement of vascular access or a CNS shunt), or significant traumatic injury within 4 weeks of the first dose of study treatment, or have an anticipated need for major surgery during the study.
5. . Presence of only leptomeningeal metastases (LM) disease confirmed by MRI and/or positive cerebrospinal fluid (CSF) pathology, with no brain metastases (BM).
6. . Prior radiation therapy for CNS metastases that involves measurable or non-measurable sites of disease to assess efficacy.
7. . Patients who have received radiation to more than 30% of the bone marrow within 2 weeks before the first dose of study treatment.
8. . Patients currently receiving (or unable to stop use at least 1 week prior to receiving the first dose of study treatment) certain medications or herbal supplements that are known to be potent inhibitors or inducers of CYP3A4/5 (see Appendix A).
9. . Unmanageable nausea and vomiting, chronic gastrointestinal diseases, or prior gastric resection or surgical procedure that may interfere with adequate absorption of study drug.
10. . History of concurrent and/or other active malignant tumors requiring treatment within 5 years of study treatment, excluding prior treated squamous cell carcinoma or basal cell carcinoma or carcinoma in situ.
11. . History of any type of documented interstitial lung disease or radiation pneumonitis.
12. . Presence of any severe or uncontrolled systemic disease or condition, including: (i) uncontrolled hypertension or diabetes; (ii) serious cardiac, pulmonary or renal disorders; (iii) active bleeding diatheses; (iv) any active type of bacterial, viral, fungal or other infection that would pose a significant risk to the patient in the opinion of the Investigator; or (v) active hepatitis B virus positive (defined as hepatitis B surface antigen (HBsAg) positive or hepatitis B core antibody (HBcAb) positive, and hepatitis B DNA positive (or detectable) or above the cut-off value) or positive HCV antibodies or positive HIV test result.
13. . Women who are pregnant or lactating. WOCBP and fertile men with a WOCBP-partner not using adequate contraception measures.
14. . Patients with unstable and symptomatic metastases: Any unstable and symptomatic CNS or distant metastasis that is not symptomatically controlled by prior surgery, radiotherapy or corticosteroid therapy within 2 weeks of initial study treatment.
15. . Any unresolved toxicities from prior therapy, greater than Common Terminology Criteria for Adverse Events (CTCAE 5.0) Grade 1 at the time of starting study treatment, with exception of alopecia.
16. . Patients with a significant cardiovascular disorder or condition, including any of the following:

    1. Congestive heart failure (CHF) currently requiring treatment and patients with New York Heart Association (NYHA) Class III/IV CHF (see Appendix B).
    2. Need for antiarrhythmic drug therapy for a ventricular arrhythmia or patients with uncontrolled or unstable arrhythmias.
    3. Severe conduction disturbance (e.g., second- or third-degree AV block).
    4. Angina pectoris requiring treatment.
    5. QTc interval > 450 msec (males) or > 470 msec (females).
    6. History of congenital long QT syndrome, congenital short QT syndrome, Torsades de Pointes, or Wolff Parkinson White syndrome.
    7. Left ventricular ejection fraction (LVEF) <50% as determined by echocardiography or MUGA scan.
    8. Myocardial infarction diagnosed within the past 6 months.
17. . Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

    1. Absolute neutrophil count <1.5 × 109/L.
    2. Platelet count <100 × 109/L (Transfusion-dependent patients are excluded from this study).
    3. Hemoglobin <90 g/L.
    4. Alanine aminotransferase (ALT) > 2.5 times the upper limit of normal (ULN) in the absence of documented metastases to liver or > 5 times the ULN in the presence of metastases to liver.
    5. Aspartate aminotransferase (AST) > 2.5 times the ULN in the absence of documented metastases to liver or > 5 times the ULN in the presence of metastases to liver.
    6. Total bilirubin > 1.5 times the ULN in the absence of metastases to liver or >3 times the ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or metastases to liver.
    7. Creatinine >1.5 times the ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft-Gault equation). Confirmation of creatinine clearance is only required when creatinine is >1.5 times the ULN.
    8. If bone metastases are present and liver function is otherwise considered adequate by the Investigator, then isolated elevated alkaline phosphatase (ALP) is not an exclusion criterion.
18. . History of hypersensitivity to active or inactive excipients of the study drug or drugs with a similar chemical structure or class to the study drug.
19. . Judgment by the Investigator that the patient should not participate in the study if the patient is unwilling to comply with all study procedures and treatment.
20. . History of recent stroke (<6 months), or prior central nervous system injury that has persistent neurologic deficits that would affect neurologic assessments.
21. . Significant medical or psychiatric illness that would interfere with the compliance to the protocol and ability to tolerate treatment.
22. . Patients who have received any anti-neoplastic herbal medicines for their malignant tumors within the past 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced non-small cell lung cancer (NSCLC) who have been diagnosed with epidermal growth factor receptor mutation type (EGFRm+) and have central nervous system (CNS) metastasis
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2031-05 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | up to 36 months
  The period from the first administration date of the study treatment to the date of death due to any cause.

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) for zorifertinib | up to 36 months
  All adverse events were classified according to the CTCAE (version: 5.0)
Incidence of Dose Adjustments for zorifertinib | up to 36 months
  The dose adjustments during the treatment by zorifertinib
Progression-free survival (PFS) | every 8 weeks,up to 36 months
  Investigator conducted the assessment based on RECIST 1.1
intracranial Progression-free survival (iPFS) | every 8 weeks,up to 36 months
  Investigator conducted the assessment based on RECIST 1.1
Objective Response Rate (ORR) | every 8 weeks, up to 36 months
  Investigator conducted the assessment based on RECIST 1.1

OTHER OUTCOMES:
The progression-free survival period of the zorifertinib treatment group (PFS2) | every 8 weeks, up to 36 months
  The period from the first administration date of the study treatment to the date of disease progression or death in the second-line treatment（Just for the zorifertinib treatment group ). Investigator conducted the assessment based on RECIST 1.1
The Genetic Resistance Status | up to 36 months
  Conduct genetic testing when disease progression occurs during the first-line zorifertinib treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu M.D., Principal Investigator — Guangdong Provincial People's Hospital
Locations (34):
- China (34):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Tumor Hospital, Beijing, Beijing Municipality
  - Capital Medical University Affiliated Beijing Chest Hospital, Beijing, Beijing Municipality
  - Chongqing University Affiliated Cancer Hospital, Chongqing, Chongqing Municipality
  - People's Liberation Army Army Specialized Medical Center, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Foshan First People's Hospital, Foshan, Guangdong
  - Heyou Hospital, Shunde District, Foshan City, Foshan, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhenzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - Nanjing Chest Hospital, Nanjing, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Dalian University of Technology Affiliated Central Hospital (Dalian Central Hospital), Dalian, Shandong
  - Qingdao University Affiliated Hospital, Qingdao, Shandong
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shenzhen Hospital, Cancer Hospital, Chinese Academy of Medical Sciences, Shenzhen, Shenzhen
  - Shenzhen Third People's Hospital, Shenzhen, Shenzhen
  - Chengdu Third People's Hospital, Chengdu, Sichuan
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Yunnan Provincial First People's Hospital, Kunming, Yunnan